CLINICAL TRIAL: NCT05741528
Title: An Open-label Extension Study to Assess the Safety and Tolerability of SEP-363856 in Subjects With Schizophrenia Switched From Typical or Atypical Antipsychotic Agents
Brief Title: An Extension Study to a Clinical Study That Will Continue to Evaluate the Effectiveness and Safety of SEP-363856 in People With Schizophrenia That Switch to SEP-363856 From Their From Their Current Antipsychotic Medication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-309
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-363856 (Experimental)
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 tablet

SUMMARY:
An Extension study to a clinical study that will continue to evaluate the effectiveness and safety of SEP-363856 in people with schizophrenia that switch to SEP-363856 from their current antipsychotic medication. This study will accept both male and female participants that have completed study SEP361-308. This study will be held in approximately 24 study sites in North America. Participation in the study will be approximately up to 25 weeks.

DETAILED DESCRIPTION:
This is a 24-week, outpatient, multicenter, flexible-dose, open-label extension study designed to evaluate the long-term safety and tolerability of SEP-363856 (50 to 100 mg/day) for the treatment of subjects with schizophrenia who have completed Study SEP361-308 treatment period, during which they were switched from a previous antipsychotic treatment to SEP-363856.

ELIGIBILITY:
Inclusion Criteria: (list is not all inclusive)

* Subject has given written informed consent and privacy authorization prior to participation in the study.
* Subject has completed the Treatment Period of Study SEP361-308.
* Subject has not taken any psychotropic medication other than the study drug, pre-switch antipsychotic and protocol-allowed medications during Study SEP361-308.
* Female subject must have a negative rapid urine pregnancy test at the End of Treatment (EOT) Visit of Study SEP361-308.

Exclusion Criteria: (list is not all inclusive)

* Subject is suicidal based on the Columbia - Suicide Severity Rating Scale (C-SSRS) assessment at the End of Treatment (EOT) Visit of Study SEP361-308.
* Subject has a clinically significant abnormality including physical examination, vital signs, or ECG finding at the End of Treatment (EOT) Visit of Study SEP361-308.
* Subject has a positive rapid urine drug screen at the EOT Visit of Study SEP361-308.
* Female subject is pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Site, Anaheim, California
  - Research Site, Bellflower, California
  - Research Site, Garden Grove, California
  - Research Site, Lemon Grove, California
  - Research Site, Santee, California
  - Research Site, Torrance, California
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Gaithersburg, Maryland
  - Research Site, Berlin, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
  Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 clinical sites in the United States (US) from 31 March 2023 to 23 September 2024.
Pre-assignment Details: A total of 75 participants rolled over from Study SEP361-308 (NCT05628103) into Study SEP361-309, and all 75 participants received at least one dose of SEP-363856 in the 24-week treatment period.
Groups:
- SEP-363856: Participants received SEP-363856 at the same dose they were taking upon completion of Study SEP361-308 (NCT05628103), orally, once daily (QD). Thereafter, the dose was adjusted within the range of 50 milligrams/day (mg/day) to 100 mg/day in 25 milligrams (mg) increments (i.e. 50 mg/day, 75 mg/day, or 100 mg/day), based on clinical judgment. Participants continued to receive flexible dose of SEP-363856 (50 mg/day to 100 mg/day) up to Week 24.
Period: Overall Study
Arm/Group | SEP-363856
Started | 75
Completed | 56
Not Completed | 19
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 2
Not completed — Non-Compliance With Study Drug | 2
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug during the 24-week open-label extension (OLE) treatment period.
Groups:
- SEP-363856: Participants received SEP-363856 at the same dose they were taking upon completion of Study SEP361-308 (NCT05628103), orally, QD. Thereafter, the dose was adjusted within the range of 50 mg/day to 100 mg/day in 25 mg increments (i.e. 50 mg/day, 75 mg/day, or 100 mg/day), based on clinical judgment. Participants continued to receive flexible dose of SEP-363856 (50 mg/day to 100 mg/day) up to Week 24.
Arm/Group | SEP-363856
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: Black or African American | 49
  Race: White | 23
  Race: Multiracial | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 13
  Ethnicity: Not Hispanic or Latino | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease occurring after the administration of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: From first dose of study drug up to end of 1 week follow up period (up to Week 25)
Population: Safety population included all participants who received at least one dose of study drug during the 24-week OLE treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 75
Participants | 28

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease occurring after the administration of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A serious adverse event is any AE occurring at any dose that results in death, is life-threatening, results in persistent or significant disability/incapacity, requires in-patient hospitalization or prolongation of existing hospitalization, or is a congenital anomaly/birth defect.
Time Frame: From first dose of study drug up to end of 1 week follow up period (up to Week 25)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 75
Participants | 4

3. Primary Outcome: Number of Participants With AEs Leading to Discontinuation of Study
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease occurring after the administration of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. AEs leading to discontinuation from the study are those AEs which caused participant to discontinue from the study.
Time Frame: From first dose of study drug up to end of 1 week follow up period (up to Week 25)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 75
Participants | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of 1 week follow up period (up to Week 25)
Description: Safety population included all participants who received at least one dose of study drug during the 24-week OLE treatment period.
Arm/Group | SEP-363856
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 4/75
Other Adverse Events (participants affected / at risk) | 9/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEP-363856 (N=75)
Delusion (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEP-363856 (N=75)
Weight decreased (Investigations) | 5
C-reactive protein increased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT05741528/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT05741528/SAP_001.pdf